CLINICAL TRIAL: NCT01179386
Title: Expectation of Driving Performance in Young Adults With ADHD Assessed by Driving Simulator and Seat Pressure Mapping
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: hermanadhd
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: methylphenidate; ADHD; driving; simulator; pressure; adolescent
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- methylphenidate: 30 adolescents who are treated with Methylphenidate will perform the driving simulator and seat pressure mapping tests, in 2 different days : 1. with their regular methylphenidate medication and 2: without the methylphenidate medication after a 4 days washout period. Results will be recorded and statistical test will be performed.
- no medication: 30 adolescents : control group , not suffering from ADHD and without methylphenidate medication will perform the driving simulator and seat pressure mapping tests. Results will be recorded and statistical test will be performed.

SUMMARY:
Adolescents suffering of ADHD may have impaired driving performance. The investigators would like to check the differences in driving performance in young adults(aged: 15-18 years) with ADHD by driving simulator and seat pressure mapping with and without methylphenidate medication.

DETAILED DESCRIPTION:
Adolescents with ADHD who are treated with one of the methylphenidate medication that is in use in Israel(Ritalin,Ritalin SR,Concerta,Ritalin LA)will be tested by driving simulator and seat pressure mapping by 2 stages: 1.when they are taking the medication that they are taking every day to control ADHD and: 2. without medication ( after 4 day washout period).

ELIGIBILITY:
Inclusion Criteria:

* age 15-18 years Suffering from ADHD treated by methylphenidate before receiving driving license

Exclusion Criteria:

* any other neurological or psychiatric problem under treatment or investment adolescents who have driving license

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 30 adolescents aged 15-18 years ,diagnosed as suffering from ADHD and being treated with a methylphenidate medication that is used in Israel 30 adolescents aged 15-18, without ADHD will the control group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: cohen he avner, md, Principal Investigator — sherute briut clalit; razon nava, Dr, Study Director — Tel Aviv University
Locations (1):
- Cohen Herman Avner, Petah Tikva, Israel

REFERENCES:
- [Background] Cox DJ, Humphrey JW, Merkel RL, Penberthy JK, Kovatchev B. Controlled-release methylphenidate improves attention during on-road driving by adolescents with attention-deficit/hyperactivity disorder. J Am Board Fam Pract. 2004 Jul-Aug;17(4):235-9. doi: 10.3122/jabfm.17.4.235. PMID 15243010